CLINICAL TRIAL: NCT04932824
Title: A Long-term Follow-up Study to the Phase 1 Study in Healthy Volunteers to Evaluate the Safety and Immunogenicity of SCB-2019, a Recombinant SARS-CoV-2 Trimeric S-Protein Subunit Vaccine for COVID-19
Brief Title: Long-term Follow-up to the Phase 1 Study of Adjuvanted SARS-CoV-2 (SCB 2019) Vaccine for COVID-19.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CLO-SCB-2019-002
Record Dates: First submitted 2021-04-13; First posted 2021-06-21 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SCB-2019 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects Without Treatment Cross-over (No Intervention): these subjects will not receive any vaccination during this study.
- Subjects With Treatment Cross-over (From 1st Dose of Active Study Vaccine Onwards) (Experimental): Once the treatment assignments of study CLO-SCB-2019-001 are unblinded, those subjects who have received placebo and provided there is active study vaccine available, will be given the option to receive 2 doses of active study vaccine 21 days apart (ie, treatment cross-over)
  Interventions: Biological: SCB-2019
- Subjects who will receive Booster Vaccine (Experimental): For subjects out of those who received SCB-2019 CpG/Alum-adjuvanted vaccine in study CLO-SCB-2019-001: the subjects will receive a booster dose.
  Interventions: Biological: SCB-2019

INTERVENTIONS:
Biological: SCB-2019 — a Recombinant SARS-CoV-2 Trimeric S-Protein Subunit Vaccine for COVID-19.
  Arms: Subjects With Treatment Cross-over (From 1st Dose of Active Study Vaccine Onwards); Subjects who will receive Booster Vaccine

SUMMARY:
To develop an effective vaccine against the Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, Clover Biopharmaceuticals is conducting a Phase 1 study (CLO-SCB-2019-001) in healthy volunteers to evaluate the safety and immunogenicity of SCB-2019, a recombinant SARS-CoV-2 trimeric Spike protein (S-protein) subunit vaccine. This study, CLO-SCB-2019-002, will be a long-term follow-up study for subjects who have completed CLO-SCB-2019-001 in order to assess longer safety and immunogenicity up to 24 months after the 1st dose of vaccination.

DETAILED DESCRIPTION:
Once a subject enrolled in the dose-escalation part of study CLO-SCB-2019-001 (groups 1-15) has completed the 6-month visit, he/she will enter this study automatically, since subjects were requested to sign the informed consent form for this long-term follow-up study at the same time they consent to study CLO-SCB-2019-001. For a subject who will receive active vaccine (subjects who received placebo in study CLO-SCB-2019-001) or a booster dose during this long-term study, an additional informed consent form will be signed prior to receiving vaccine.

After study CLO-SCB-2019-001 ends and the treatment assignments are unblinded, those subjects who have received placebo will be given the option to receive 2 doses of active study vaccine 21 days apart (defined as treatment cross-over); subjects who do not consent to vaccination will be discontinued from the study. Subjects who consent to vaccination will be followed up until 18 months after the 1st dose of the cross-over vaccination.

Subjects that received SCB-2019 vaccine adjuvanted with AS03 in study CLO-SCB-2019-001 will be followed up for safety only for 12 months after the 1st dose received (V10, day 366).

Of the subjects that received SCB-2019 CpG/Alum-adjuvanted vaccine in study CLO-SCB-2019-001, the first 24 subjects that agree to receive booster dose will be consented to an additional informed consent form prior to receiving a booster dose and included in this long-term follow-up study. These 24 subjects will be followed up until 12 months after the booster dose.

Statistical methods:

The following descriptive statistics will be used as applicable to summarize the study data unless otherwise specified. Individual subject data will be presented in listings.

* Continuous variables: sample size [n], mean, standard deviation [SD], median, minimum [Min], and maximum [Max].
* Categorical variables: frequencies and percentages. All safety analyses will be performed on the Safety Analysis Set. Adverse events will be coded using Medical Dictionary for Regulatory Activities (MedDRA) central coding dictionary, version 22.0 (or higher). The percentage of subjects with at least 1 adverse event (AE), adverse event of special interest (AESI), or serious adverse event (SAE) will be tabulated with exact 95% confidence interval (CI) for each treatment and overall. Adverse events/SAEs leading to withdrawal and all pregnancies occurring during the study period will be tabulated with exact 95% CI. The percentage of subjects with at least 1 local AE (solicited and unsolicited), at least 1 general AE (solicited and unsolicited) and any AE will be tabulated, with exact 95% CI. The same computations will be done for Grade 3, any AEs considered related to vaccination, any Grade 3 AEs considered related to vaccination, SAEs and AESIs. Analysis of immunogenicity will be based on the Per Protocol Set. If, at any timepoint, the percentage of vaccinated subjects with serological results excluded from the Per Protocol Set for analysis of immunogenicity is 10% or more, a second analysis based on the Immunogenicity Analysis Set will be performed to complement the Per Protocol Analysis. Observed values and ratio/change from Baseline values (as applicable) will be summarized for each treatment (placebo, vaccine, and with addition of each adjuvant) and at each timepoint where blood samples are collected. Individual data listings of any Coronavirus disease 2019 (COVID-19) cases during the study will be provided. Number of cases that undergo COVID-19 workup as well as the incidence of COVID-19 positive results will be individually listed and summarized using summary statistics per treatment group and per protocol scheduled time point. Time to COVID-19 positive result will also be summarized using Kaplan-Meier methods and the median time to COVID-19 positive result will be estimated and presented with the 95% CIs, if estimable, separately for each treatment group. In addition, clinical risk assessment of COVID-19 at the time of the case workup as assessed by the National Early Warning Score 2 (NEWS2) system will be individually listed and summarized per treatment group.

ELIGIBILITY:
Inclusion Criteria:

* All subjects from study CLO-SCB-2019-001 will automatically move on to this long-term follow-up study if: 1) They have given informed consent for this follow-up study; and 2) They have completed the D184 visit of study CLO-SCB-2019-001 (ie, 6 months post the 1 st vaccination).

Exclusion Criteria:

* All subjects who did not participate and completed the study or did not signed the inform consent for this follow up study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Incidence of AESIs and SAEs | from 6 to 24 months after the 1st vaccination dose
  To evaluate the safety profile of SCB-2019 up to 24 months after the 1st vaccination dose
Incidence of AESIs and SAEs | up to 12 months after booster dose
  To evaluate the safety profile of SCB-2019 up to 12 months after booster dose
Serum anti-SCB-2019 IgG antibody titers | from 6 to 24 months after the 1st vaccination dose
  To describe and compare antibody response kinetics in response to vaccination with SCB-2019 up to 24 months after the 1st vaccination dose
Serum anti-SCB-2019 IgG antibody titers | up to 12 months after booster dose
  To describe and compare antibody response kinetics in response to vaccination with SCB-2019 up to 12 months after booster dose

SECONDARY OUTCOMES:
Serum anti-SARS-CoV-2 neutralizing antibody titers (ACE2 receptor-based) | from 6 to 24 months after the 1st vaccination dose
  To describe serum immune responses in terms of antibody titers competitive with binding to ACE2
Serum anti-SARS-CoV-2 neutralizing antibody titers (ACE2 receptor-based) | up to 12 months after booster dose
  To describe serum immune responses in terms of antibody titers competitive with binding to ACE2

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Nedlands, Territory Western Australia, Australia